CLINICAL TRIAL: NCT03023644
Title: Improving Neurodevelopmental Outcomes in Children With Congenital Heart Disease: An Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jane W. Newburger, MD, MPH, Commonwealth Professor of Pediatrics, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB-P00022440
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Congenital Heart Defect; Executive Function; Children; Neurodevelopmental Disorders; Working Memory; Infant Open Heart Surgery
Keywords: Congenital Heart Disease; Neurodevelopmental Disorders; Children; Executive Function; Working Memory; Cognitive interventions; Infant Open Heart Surgery
MeSH Terms: conditions — Heart Defects, Congenital; Neurodevelopmental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cogmed Working Memory Training (Experimental): The group randomized to the intervention will receive Cogmed computerized training of executive function and attention skills. The standard Cogmed RM will be used for this trial arm. This is a child-friendly web-based software program. The investigators will use a version of the program that contains 12 different neurocognitive tasks. Tasks become more difficult as a function of performance on a session-by-session basis. Each training session lasts 35-40 minutes, with one session to be completed per day 5 days each week for 5 weeks, for a total of 25 sessions. The program yields individual session-by-session and task-by- task training results, including the children's responses, time spent on each task, and evolution curves.
  Interventions: Behavioral: Cogmed Working Memory Training
- Standard of Care (No Intervention): Children randomly assigned to the control group will receive the standard of care recommended for patients with critical CHD. This includes cardiac surveillance and neurodevelopmental counseling and screening at our Cardiac Neurodevelopmental Program if needed. Once enrolled in our study, a child in the control group will not receive Cogmed intervention or any other cognitive intervention that targets executive functions or ADHD symptoms until after the 3-month follow-up neurodevelopmental evaluation is performed, i.e., 5-6 months after initial enrollment. Like children assigned to the intervention group, controls can continue on treatments that are already in place for other neurodevelopmental disabilities (e.g., speech therapy, occupational services).

INTERVENTIONS:
Behavioral: Cogmed Working Memory Training — Cogmed Working Memory Program will be used as a computerized home-based intervention. Families will an iPad with a web-based software program. The 25 sessions will be completed individually by the child with parental supervision. For the first 5 sessions, the participant trains on the same set of games; on the 6th session and every 5th session thereafter, a new task is introduced and replaces one of the initial tasks. At the end of each session, the child can play an age-appropriate computerized game as a reward. After each session, results are uploaded by parents to a secure website, to keep track of the participant's progress. Families will be contacted weekly to check program function and discuss concerns.
  Arms: Cogmed Working Memory Training

SUMMARY:
Each year, approximately 1 child in every 100 is born with Congenital Heart Disease (CHD), making it the most common birth defect. With recent medical advances, more children with CHD survive early open-heart surgery, so that there are now 2 to 3 million adult survivors with CHD. These survivors face challenges in terms of their cognitive and behavioral development. For many, the limitations affect their academic achievement, social adaption and, ultimately, their quality of life. Among the most disabling limitations are those that pertain to the ability to maintain attention, plan and organize activities, regulate emotions, and develop problem-solving strategies. Collectively, these are referred to as executive functions (EF) because they are higher-order abilities that enable one to coordinate complex behaviors. Additionally, impaired EF also underlie mental health disorders. In spite of the abundance of evidence that children with CHD struggle with EF, there is little to offer them in the way of evidence-based interventions to prevent or mitigate these problems.

The investigators propose to conduct the first randomized trial to evaluate the efficacy of an intervention, the Cogmed Working Memory Program, in improving the neurodevelopment outcomes of children with critical CHD after infant open-heart surgery. Children who meet eligibility criteria and who agree to participate will be randomly assigned to an intervention or control group. Children in the intervention group will complete 25 35-40 minute sessions of Cogmed training, spread over for 5 weeks. This Program is a set of home-based, child-friendly, computerized activities. The control group will receive the standard of care for children with CHD. Children's scores on EF and related neurodevelopmental tests will be evaluated before the intervention group completes Cogmed training, at the conclusion of their training, and 3 months later. The latter assessment will indicate whether any gains in EF skills of the children in the intervention group are sustained after training. Parents and teachers will also complete questionnaires about children's EF, attention, and social behaviors to determine whether training affects behaviors of the intervention group at home and in school. The investigators will also identify the medical and surgical characteristics of children who benefit most from Cogmed training. This information will be helpful in targeting the intervention most efficiently in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Open heart surgery before age 12 months of life
2. Ages between 7 years 0 months and 12 years 11 months
3. ≥6 months post-cardiac surgery at enrollment
4. Cardiology follow-up (clinic or inpatient) at BCH or other affiliated center in the last 6 years.
5. English and/or Spanish speaking
6. Informed consent of parent/guardian as well as assent of child

Exclusion Criteria:

1. Known chromosomal anomalies and/or genetic syndromes
2. Severe physical and/or sensory impairments (hearing, visual, or psychomotor) that would prevent use of the computerized program and tablets
3. Confirmed formal diagnosis of any autism spectrum disorder or a severe developmental and/or intellectual disorder that would prevent successful completion of the planned study testing.
4. Scheduled to undergo major cardiac interventions in the 6 months following enrollment
5. Received, receiving, or scheduled to receive Cogmed or any other computerized behavioral training program targeting executive functions or ADHD

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline scores at the computerized Working Memory Test from the NIH Toolbox Assessment of Neurological and Behavioral Function at post-treatment assessment | 2 weeks
  This standardized measure assesses the ability to process information across a series of modalities (visual-spatial and verbal), to hold this information in a short-term buffer, and to actively manipulate it mentally. It is considered an excellent composite indicator of children's executive function skills, as it requires the simultaneous implementation of control of attention and working memory abilities on tasks of increasing complexity. Mean scores are automatically computed and are compared to a standardization sample of US children of the same age. They are normally distributed (mean=100, SD=15).

CONTACTS AND LOCATIONS:
Overall Officials: Jane W Newburger, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share the final research data, including the computerized dataset upon which publications were based. The final dataset may also include both raw data and derived variables. Data products from this study will be made available without cost to researchers and analysts. User registration will be required in order to access or download files. As part of the registration process, users must agree to the conditions of use governing access to the public release data, including restrictions against attempting to identify study participants, destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistribution of the data to third parties, and proper acknowledgement of the data resource. We are aware of the need to protect human subject information and Protected Health Information in accordance with HIPPA standards and in other situations where data sharing may not be appropriate or allowed. Data sharing will occur in a timely fashion.

REFERENCES:
- [Derived] Calderon J, Bellinger DC, Hartigan C, Lord A, Stopp C, Wypij D, Newburger JW. Improving neurodevelopmental outcomes in children with congenital heart disease: protocol for a randomised controlled trial of working memory training. BMJ Open. 2019 Feb 19;9(2):e023304. doi: 10.1136/bmjopen-2018-023304. PMID 30782877